CLINICAL TRIAL: NCT02775227
Title: HYPAR Trial - Hydrocortisone vs Pasireotide in Reducing Pancreatic Fistula and Other Complications After Pancreatic Resection - a Prospective, Randomized, Controlled Trial
Brief Title: HYPAR Trial - Hydrocortisone vs. Pasireotide in Reducing Pancreatic Surgery Complications
Acronym: HYPAR
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Ville Sallinen, MD, PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: HYKS-190116
Record Dates: First submitted 2016-05-14; First posted 2016-05-17 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Pancreatic Fistula; Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Fistula; Pancreatic Neoplasms | interventions — Hydrocortisone; pasireotide

ARMS (2):
- Hydrocortisone (Experimental)
  Interventions: Drug: Hydrocortisone
- Pasireotide (Active Comparator)
  Interventions: Drug: Pasireotide

INTERVENTIONS:
Drug: Hydrocortisone
  Arms: Hydrocortisone
Drug: Pasireotide
  Arms: Pasireotide

SUMMARY:
Pancreatic resections carry a high risk for complications, especially pancreatic fistula. Both hydrocortisone and pasireotide have been shown to be effective in reducing complications in earlier RCTs. The aim of this study is to compare the effectiveness and safety of these two drugs in preventing complications of pancreatic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for pancreatic surgery (pancreaticoduodenectomy, distal pancreatectomy, enucleation, or other type of pancreatic resection)

Exclusion Criteria:

* Preoperative exclusion criteria:
* Atrophic pancreas and/or dilated pancreatic duct at the site of planned pancreatic transsection (applies only to patients undergoing pancreaticoduodenectomy)
* Total pancreatectomy planned
* Allergy or other contraindication for hydrocortisone or pasireotide
* Age < 18 years
* No informed consent
* Intraoperative exclusion criteria:
* Pancreatic resection cancelled (e.g. disseminated cancer)
* Hard pancreas and/or dilated pancreatic duct discovered during operation (applies only to patients undergoing pancreaticoduodenectomy)
* Total pancreatectomy is performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Complication Index | 30 days postoperatively

SECONDARY OUTCOMES:
Complications (Clavien-Dindo classification) | 30 days postoperatively
Postoperative pancreatic fistula (ISGPS-classification) | 30 days postoperatively
Postoperative delayed gastric emptying (ISGPS-classification) | 30 days postoperatively
Post-pancreatectomy hemorrhage (ISGPS-classification) | 30 days postoperatively
Length of hospital stay, days | During hospital stay, on average 7-14 days
Readmissions | 30 days postoperatively

OTHER OUTCOMES:
Number of patients receiving adjuvant therapy | 6 months postoperatively
Overall survival | 10 years
Disease free survival | 10 years
Disease specific survival | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Derived] Tarvainen T, Siren J, Kokkola A, Sallinen V. Effect of Hydrocortisone vs Pasireotide on Pancreatic Surgery Complications in Patients With High Risk of Pancreatic Fistula: A Randomized Clinical Trial. JAMA Surg. 2020 Apr 1;155(4):291-298. doi: 10.1001/jamasurg.2019.6019. PMID 32022887